CLINICAL TRIAL: NCT00123838
Title: Beacon® Transponder Implantation and Localization in the Prostate
Brief Title: Positioning and Tracking the Prostate During External Beam Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prostate Stage 3
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Radiotherapy; Neoplasm; Localization; Tracking; Cancer of Prostate; Neoplasms, Prostate
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group Assignment (Experimental): Calypso® 4D Localization System
  Interventions: Device: Calypso® 4D Localization System

INTERVENTIONS:
Device: Calypso® 4D Localization System — Localization of prostate irradiation.

SUMMARY:
The purpose of this study is to evaluate a non-ionizing electromagnetic method to align the prostate treatment site for radiation therapy and to monitor its position throughout radiation therapy delivery. The clinical study involves using an investigational device, the Calypso® 4D Localization System, and requires permanent implantation of three small sensors called Beacon® transponders in the prostate.

DETAILED DESCRIPTION:
The goal for prostate radiation therapy is to give a high dose of radiation to the prostate and a minimal dose to the healthy tissue around the prostate. It is well known that the prostate moves slightly within the pelvis and that its position varies a few millimeters from day to day. There are several methods used to position the body and the prostate accurately at the beginning of each radiation therapy session.

One of the standard methods is to permanently implant small markers (gold spheres or cylinders) in the prostate and use x-rays in the radiation therapy treatment room to determine whether the markers are in the correct position. If the markers are in the correct position, then the assumption is that the prostate also is in the correct position. If the markers are not in the correct position on the x-ray, then the table that the patient lies on can be shifted so that the markers are in the right place.

In this study the Beacon® transponder will be used in place of the standard gold marker. During the radiation therapy visits, the patient position in the treatment room will be corrected using the Beacon transponder with an investigational system, called the Calypso® 4D Localization System. The Calypso system consists of a flat panel, placed over the pelvis and connected to a computer, which monitors the position of the Beacon transponders within the prostate. During five radiation therapy appointments and one extra visit, the position of the markers in the prostate will be confirmed with x-rays.

The Beacon transponder is a small glass cylinder that contains a tiny electrical circuit. The glass vial is completely sealed and separates the internal components (i.e., the electrical circuit) from the rest of the body. The glass vial is approximately one-third of one inch long and one-tenth of one inch in diameter. Three Beacon transponders will be implanted in the prostate. They will be permanently implanted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed diagnosis of prostate cancer
* Intact prostate (minor transurethral resection of the prostate [TURP] defects are allowed at the discretion of the investigator)
* Ability to comply with study visit schedule

Exclusion Criteria:

* Prior treatment for prostate cancer.
* Prostate cancer stage IV (metastatic disease).
* Patients who are not eligible for prostate biopsy.
* Past history of abdominoperineal (A-P) resection.
* Planned course of treatment using brachytherapy (permanent brachytherapy seeds or high dose rate [HDR] brachytherapy).
* Allergy to local anesthetics.
* Patients with any permanently implanted medical devices that have an energy source, such as pacemakers, defibrillators, neurostimulators, and drug infusion pumps; this also includes prosthetic implants in the abdomen or pelvis, such as an artificial hip; or vascular implants such as arterial stents or stent-grafts for aortic aneurysms. This does not include surgical clips, staples or coronary stents.
* History of chronic prostatitis.
* Patients with a history of recent acute and/or chronic bleeding disorders.
* Patients on therapeutic anti-coagulants or anti-platelet therapy, not including aspirin.
* Patients for which the maximum anterior-posterior separation through the torso minus the height of the center of the prostate is greater than 23 cm. (Measurements will be made visually with a ruler.)
* Baseline evaluation shows an INR or PTT outside of the normal range for the institution; platelet count < 75,000 mm3; or creatinine > 2.0 mg/dl.
* Any other medical condition or laboratory value that would, at the discretion of the investigator, preclude the patient from participation in a clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Radiographic verification of at least five of approximately 40 radiation treatment days | 8 weeks

SECONDARY OUTCOMES:
Patient Preference Questionnaire and SF 36 Health Survey at five radiation treatment days | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Levine, Ph.D., Study Director — Varian, a Siemens Healthineers Company
Locations (5):
- United States (5):
  - Scottsdale Healthcare - Osborn, Scottsdale, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - The Nebraska Medical Center, Omaha, Nebraska
  - The Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No